CLINICAL TRIAL: NCT04343807
Title: Effectiveness of Ultrasound Guided PECS Block on Opioid Consumption and Patient Satisfaction Through Adequate Pain Control Following Breast Cancer Surgery. A Prospective Randomized Controlled Trial
Brief Title: Effectiveness of Ultrasound Guided PECS Block on Opioid Consumption and Patient Satisfaction Through Adequate Pain Control Following Breast Cancer Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Faisal Shamim, Associate Professor Anaesthesiology, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3543
Record Dates: First submitted 2020-04-10; First posted 2020-04-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm Female; Pain, Postoperative; Pain; Analgesia; Anaesthesia; Breast Cancer
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia; Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS block (Active Comparator): For patients in PECS group (PG), after induction of general anesthesia, the nerve block will be performed using the ultrasound-guided technique described by Blanco and colleagues. Block will be performed with a 22-gauge 100 mm needle (Stimuplex, B. Braun Medical Inc., Pennsylvania, USA) using Mindray M7 imaging system (Diagnostic Instruments Inc., China) with a high-frequency (6-13 MHz) linear array transducer.20 mL of ropivacaine 0.25% in 5-mL increments will be injected, aspirating gently between injections. The needle will be withdrawn to place the tip in the fascial plane between the pectoralis major and pectoralis minor muscles and ropivacaine 0.25%, 10 ml in 5 ml increments will be injected. Injectate spread between the muscles will be visualized. For patients in control group, no nerve block will be performed and only intravenous nalbuphine will be given.
  Interventions: Procedure: PECS Block
- Control Group (Active Comparator): For patients in control group, after induction of general anesthesia, no nerve block will be performed and only intravenous nalbuphine will be given.
  Interventions: Other: Control Group

INTERVENTIONS:
Procedure: PECS Block — PECS nerve block will be performed using the ultrasound-guided technique described by Blanco and colleagues. Block will be performed with a 22-gauge 100 mm needle (Stimuplex, B. Braun Medical Inc., Pennsylvania, USA) using Mindray M7 imaging system (Diagnostic Instruments Inc., China) with a high-frequency (6-13 MHz) linear array transducer.20 mL of ropivacaine 0.25% in 5-mL increments will be injected, aspirating gently between injections. The needle will be withdrawn to place the tip in the fascial plane between the pectoralis major and pectoralis minor muscles and ropivacaine 0.25%, 10 ml in 5 ml increments will be injected. Injectate spread between the muscles will be visualized. For patients in control group, no nerve block will be performed and only intravenous nalbuphine will be given.
  Arms: PECS block
Other: Control Group — No nerve block will be performed and only intravenous nalbuphine will be given.
  Arms: Control Group

SUMMARY:
Breast cancer is the most common and leading cause of cancer deaths among females worldwide. Patients undergoing modified radical mastectomy (MRM) are associated with moderate to severe acute postoperative pain and shoulder mobility restriction.

This study aims to determine the effectiveness of ultrasound-guided PECS block for reducing opioid consumption, providing adequate postoperative pain management and improving patient satisfaction following breast cancer surgery.

DETAILED DESCRIPTION:
The traditional pain management for patients undergoing MRM has relied heavily on opioids but a number of multimodal pain control strategies also exist including combining opioids with NSAIDs, cyclooxygenase-2 inhibitors, acetaminophen and regional blocks. Recently, literature underlines the importance of performing regional anaesthetic and analgesic techniques for postoperative analgesia following breast surgery. PECS (Pectoral nerve block) block provides analgesia for breast surgeries with few adverse effects.

OBJECTIVES To evaluate the effect of ultrasound guided pectoral block in reducing intraoperative and postoperative opioid consumption following modified radical mastectomy.

The secondary objective is to determine patient satisfaction levels associated with adequate pain control.

HYPOTHESIS Pectoral nerve blocks provides superior analgesia with less opioid consumption and improves patient satisfaction in postoperative period compared to conventional pain management for modified radical mastectomy patients

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective modified radical mastectomy (MRM)
* All adults aged between 18 and 65 years
* ASA (American Society of Anesthesiologists ) I & II

Exclusion Criteria:

* Patient refusal
* Hypersensitivity to local anaesthetics
* Coagulopathy or bleeding diathesis
* Local infection at the site of block
* BMI more than 35 kg/m2
* Chest wall deformity or previous breast surgery
* MRM with latissimus dorsi or deep inferior epigastric perforator flap reconstruction

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Total intraoperative opioid consumption | During surgical procedure
  Total intraoperative nalbuphine
Total postoperative opioid consumption | First 24 hours after surgery
  Total Rescue Tramadol Consumption

SECONDARY OUTCOMES:
Patient Satisfaction | First 24 hours after surgery
  Patient satisfaction with post-operative analgesia will be noted via satisfaction scoring i.e.:
  1. = Not Satisfied
  2. = Good or satisfied
  3. = Excellent or very satisfied
Postoperative pain score | 1, 6,12 and 24 hours after surgery
  Numeric rating scale for pain assessment: Patient will be asked to rate their intensity of pain on numeric scale from 0 (no pain) to 10 (worst possible pain).
Postoperative nausea and vomiting | First 24 hours after surgery
  Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Shamim, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] M N, Pandey RK, Sharma A, Darlong V, Punj J, Sinha R, Singh PM, Hamshi N, Garg R, Chandralekha C, Srivastava A. Pectoral nerve blocks to improve analgesia after breast cancer surgery: A prospective, randomized and controlled trial. J Clin Anesth. 2018 Mar;45:12-17. doi: 10.1016/j.jclinane.2017.11.027. Epub 2017 Dec 11. PMID 29241077
- [Background] Morioka H, Kamiya Y, Yoshida T, Baba H. Pectoral nerve block combined with general anesthesia for breast cancer surgery: a retrospective comparison. JA Clin Rep. 2015;1(1):15. doi: 10.1186/s40981-015-0018-1. Epub 2015 Sep 23. PMID 29497647